CLINICAL TRIAL: NCT07198880
Title: Impact of Home Non Invasive Ventilation in Patients With Chronic Obstructive Pulmonary Disease Discharged From Assiut University Hospital
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Mahmoud Ahmed AbdAllah, Principal investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NIV in COPD Patients
Record Dates: First submitted 2025-09-14; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: COPD; COPD (Chronic Obstructive Pulmonary Disease); Ventilation Therapy; Non Invasive Ventilation (NIV); BiPAP; Hypercapnia; Long Term Oxygen Therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypercapnia | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIV Group (Experimental): Patients who can afford to buy or attain a Bi-PAP device will be enrolled in this interventional group long-term NIV (Bi-PAP), They will also keep taking their optimal medical therapy, with or without LTOT according to oxygen status.
  Interventions: Device: BiPAP device (non invasive ventilation); Drug: Optimal Medical Management ( long acting beta agonist , long acting muscarinic antagonist and inhaled corticosteroids)
- Control Group (Active Comparator): Patients who cannot attain a BiPAP device are managed with their optimal medical therapy, with or without LTOT according to oxygen status
  Interventions: Drug: Optimal Medical Management ( long acting beta agonist , long acting muscarinic antagonist and inhaled corticosteroids)

INTERVENTIONS:
Device: BiPAP device (non invasive ventilation) — BiPAP initiated 2-4 weeks post-discharge; IPAP 16 cmH₂O (titrate), EPAP 4 cmH₂O; supplemental O₂ as needed monitor SpO₂, ABG, vitals; target ≥20% PaCO₂ reduction, improved pH, reduced work of breathing; adherence ≥4 hrs/nigh
  Scheduled monitoring of SpO₂, symptoms, and adherence; outpatient follow-up at 2-4 weeks and after 1, 3, 6 ,12 month intervals
  Arms: NIV Group
Drug: Optimal Medical Management ( long acting beta agonist , long acting muscarinic antagonist and inhaled corticosteroids) — Patients will continue on standard COPD management: inhaled bronchodilators, inhaled corticosteroids, LTOT when required, but without NIV

SUMMARY:
This study aims to evaluate the impact of long-term home non-invasive ventilation (NIV) on patients with COPD

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major cause of morbidity and mortality worldwide . A subset of patients develops chronic hypercapnia, which is linked to frequent hospitalizations, reduced quality of life, and poor survival. Despite optimized pharmacological therapy, pulmonary rehabilitation, and long-term oxygen therapy (LTOT), outcomes in these patients remain unsatisfactory.

Early randomized trials failed to show survival benefit from home Non Invasive Ventilation , largely due to low ventilatory pressures, poor adherence, and heterogeneous patient selection . More recent studies suggest a positive impact and demonstrated improved long-term survival, some studies reported reduced mortality with high-intensity NIV targeting PaCO₂ reduction .

Meta-analyses indicate that patients with persistent hypercapnia after an acute exacerbation are most likely to benefit , though uncertainties remain regarding patient selection and long-term real-world outcomes.

Management of chronic hypercapnic COPD currently includes pharmacological treatment, LTOT, and rehabilitation.

NIV is a cornerstone in acute exacerbations, but its role in the chronic setting is not universally established, and routine use in home care is limited.

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 18 year old.
* Severe COPD (classified as GOLD stage Ⅲ and IV), confirmed by FEV₁/FVC < 70% and FEV₁ < 50% of the predicted value. (9)
* Persistent hypercapnia (PaCO₂ ≥ 60 mmHg ≥2 weeks after resolution of acute exacerbation and compliant on optimal medical therapy with or without long term oxygen therapy

Exclusion Criteria:

* Other significant respiratory disorders (e.g,history suggestive OSA, Body Mass Index more than 30, pneumothorax, bullous lung disease, advanced interstitial lung diseases , restrictive thoracic wall diseases , neuromuscular disease).
* Undergone intubation or tracheostomy prior to NIV initiation during the last 2 months.
* Those using addictive narcotic medications.
* Comorbidities and diseases that might confound survival outcomes (e.g., malignancy, advanced hepatic or renal diseases).
* Pregnancy
* Refusal or Inability to tolerate NIV during initiation and adaptation phase.
* Expected Poor compliance (patients deemed unlikely to adhere to nightly NIV use such as no family support, severe frailty).
* Withdrawal criteria: stopping bipap or medical treatment, voluntary withdrawal by the participant, failure to attend scheduled visits, and significant clinical deterioration requiring alternative management during the study period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in arterial blood gas parameter "PaCO₂" | 1 year
  follow up PaCo2 level measured by mmhg
Assessment of Adherence to BiPAP therapy | 1 year
  measured as the average hours of nightly use

SECONDARY OUTCOMES:
Improvements in quality of life | 1 year
  Measured using the validated St. George's Respiratory Questionnaire - COPD. Scale range: 0-100 (0 = no impairment, 100 = maximum impairment). Direction: Higher scores indicate worse quality of life.
Improvement in Dyspnea | 1 year
  Measured using the Modified Medical Research Council (mMRC) Dyspnea Scale. Scale range: 0-4 (0 = no breathlessness, 4 = severe breathlessness). Direction: Higher scores indicate worse dyspnea.
Improvement in COPD-Related Symptoms | 1 year
  Measured using the COPD Assessment Test (CAT). Scale range: 0-40 (0 = no symptoms, 40 = very severe symptoms). Direction: Higher scores indicate more severe symptoms and worse impact on daily life.
Total Duration of COPD-Related Hospitalization per Year | 1 year
  Documented as the cumulative number of days spent in hospital for COPD exacerbations during the study period.
  Unit of Measure: Days hospitalized per participant per year
Number of COPD-Related Hospitalizations per Year | 1 year
  Documented as the total number of hospital admissions for COPD exacerbations during the study period.
  Unit of Measure: Number of hospitalizations per participant per year
Assessment of Overall survival | 1 year
  Assessment of Overall survival between 2 cohorts (one year mortality)